CLINICAL TRIAL: NCT03186105
Title: Evaluation of the Ambulatory Feasibility of Appendicectomy for Acute Appendicitis in Children 6 to 17 Years
Brief Title: Feasability of Ambulatory Appendicectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-HPNCL-05
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2018-07

CONDITIONS: Appendicitis Acute
Keywords: Appendicitis Acute; AMBULATORY
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ambulatory appendicectomy (Experimental): The intervention consist of an ambulatory care by appendicectomy of the acute appendicitis. The normal care is an appendicectomy and an hospitalisation during 2 or 3 days.
  Interventions: Other: Ambulatory appendicectomy

INTERVENTIONS:
Other: Ambulatory appendicectomy — The intervention consist of an ambulatory care by appendicectomy of the acute appendicitis. The normal care is an appendicectomy and an hospitalisation during 2 or 3 days .

SUMMARY:
The investigators will conduct a monocentric prospective preliminary study evaluating the feasibility of appendectomy for simple acute appendicitis in a cohort of 6-17 year-old children presenting to the emergency department of the Hôpital Pédiatrique de Nice CHU-Lenval (Lenval Childre Hospital, Nice) on a Period of 1 year.

DETAILED DESCRIPTION:
Acute appendicitis represents the first visceral surgical emergency of the child in terms of frequency, resulting in hospitalization, hospitalization and family costs, as well as an alteration in family dynamics.

Reducing the duration of hospitalization and allowing the child to return more quickly to his usual environment would not only reduce the risks of nosocomial infections and the workload of medical and paramedical teams but would reduce the emotional burden for the child, In addition to its consequences in terms of professional disorganization induced in the parents by the hospitalization of their child. Ambulatory hospitalization would also reduce the cost of this pathology.

In the context of ambulatory surgery, the patient's journey from admission to hospital must be perfectly codified; The novelty of this study lies in the fact of applying this mode of hospitalization to emergency surgery.

Once the consultation for abdominal pain by an emergency pediatrician carried out, the diagnostic orientation is confirmed by a visceral pediatric surgeon who performs a biological check-up and an abdominal ultrasound. After confirmation of eligibility for ambulatory care according to national recommendations and informed consent, the child is - according to the time of care and the clinical condition of the patient - immediately hospitalized in the unit (UCA) be allowed to return to his home with reconviction in the ambulatory surgery unit the next morning, at the opening of the service, on an empty stomach.

The abdominal ultrasound confirms the orientation and the diagnosis of acute appendicitis simple is posed.

The laparoscopic appendectomy is performed after the anesthesia consultation. The patient is monitored and replenished early in the UCA according to a standardized and computerized protocol.

The return home is authorized by the confirmation of "aptitude to the street" by systematic consultation of a senior surgeon and an anesthetist.

The surgical and anesthetic techniques remain the same as in traditional surgery, but the timing is organized for an outpatient treatment The follow-up of the child will be carried out as early as day 1 by the call of the UCA, then at day 8 during postoperative consultation and finally at day 30 post-operative per call.

ELIGIBILITY:
Inclusion Criteria:

* Boy or girl
* Subjects aged 6 to 17 years (Children under 6 years of age with a table of acute appendicitis will not be included in the high probability of complicated acute appendicitis in these young children who are often rapidly changing pathology or delayed diagnosis Patients over 17 years of age are usually referred to adult hospitals and will not be included)
* Surgical indication of appendectomy under laparoscopy for simple acute appendicitis according to clinico-biological criteria (Appendix 6).
* Ambulatory eligibility according to the criteria usually defined
* Dosage of negative bHCG (exclusion of pregnancy)
* Parents and children able to understand the study and having signed informed consent
* Possibility of organizing childcare immediately at home
* Subjects and holders of parental authority who have given their informed and written consent
* Subjects affiliated to Social Security system

Exclusion Criteria:

* Patients who had spent an overnight stay in hospital prior to surgery and therefore could not meet the ambulatory criteria.
* An ASA score higher than III
* Impossibility of ambulatory surgery due to a residence outside the coverage area defined by the surgical and ambulatory anesthesia service, the impossibility of being transported after returning home, the absence of parents Child after discharge from hospital
* Contra-indication to the practice of an appendectomy under laparoscopy

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-06-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of ambulatory care | day 8 after intervention
  Feasibility is defined as the association of the return to the patient's home within the twelve hours of the intervention and the absence of re-hospitalization or recourse to town medicine before the postoperative consultation at day 8

SECONDARY OUTCOMES:
pain of the patient at home | 3 post-operative days
  To evaluate pain in the home, parents will be given a heterogeneous questionnaire in the form of a grid represented by a validated tool evaluating the management of the pain on the 3 post-operative days. PPMP Scale (Postoperative Pain Measure for Parents )
rate of patients able to return home on the day of the intervention | the day of the intervention at day 0
  pediatric postanesthetic discharge scoring system (Ped-PADSS) ≥ 9 / 10
rate of consultations at Emergencies unit care before 8 days post operative | 8 days post operative
  Evaluation through study of files on computer server of the Emergencies unit care before 8 days post operative
Parent Satisfaction | 8 days post operative
  Parent Satisfaction will be assessed through a questionnaire
Patient Satisfaction | 8 days post operative
  Patient Satisfaction will be assessed through a questionnaire
number of overnight stays caused by the failures of ambulatory care | 8 days post operative
  All hospitalization nights will be counted for patients in check up to day 8 in immediate postoperative
re-admission rate at day 30 | 30 days post operative
  The readmission rate will be defined as the percentage of patients rehospitalized at least once to 30 days for specific complications of the intervention or appendicitis.
the rate of fallback due to specific complications of the intervention or appendicitis | the day of the intervention at day 0
  The fallback rate is defined by the ratio of the number of patients transferred in conventional surgery to the total number of patients included in the study and operated
Parental satisfaction 1 day post operative | 1 day post operative
  Parent Satisfaction will be assessed by a Likert scale which will be proposed during a telephone call
Parental satisfaction 30 days post operative | 30 days post operative
  Parent Satisfaction will be assessed by a Likert scale which will be proposed during a telephone call

CONTACTS AND LOCATIONS:
Overall Officials: Florence BASTIANI, MD, Principal Investigator — Hôpitaux Pédiatriques de Nice CHU-LENVAL
Locations (1):
- Hôpitaux Pédiatriques de Nice CHU-LENVAL, Nice, France

IPD SHARING:
Plan to Share IPD: No